CLINICAL TRIAL: NCT04856579
Title: Assessment of Seminal Levels of Cystatin C and Endoglin in Infertile Men With Varicocele
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Essam Mohamed El-sayed Akl, Assistant Professor, Benha University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RC-5-4-2021
Record Dates: First submitted 2021-04-06; First posted 2021-04-23 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Varicocele; Infertility, Male
Keywords: Male infertility; Varicocele; Cystatin C; Endoglin
MeSH Terms: conditions — Varicocele; Infertility, Male

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Varicocelectomy (Other): Subinguinal varicocelectomy under general anesthesia and complete aseptic condition
  Interventions: Procedure: Varicocelectomy

INTERVENTIONS:
Procedure: Varicocelectomy — Subinguinal varicocelectomy under general anesthesia and complete aseptic condition

SUMMARY:
Varicocele is a major contributor in male infertility. The improvement of sperm parameters after varicocelectomy supports this contribution. The pathophysiological mechanisms of varicocele-induced male infertility are still under investigation. Cystatin C (Cys C) and endoglin are secreted glycoproteins that recently linked to several cellular changes common in varicocele like apoptosis and autophagy.

DETAILED DESCRIPTION:
Subinguinal varicocelectomy under general anesthesia and complete aseptic condition was done to infertile men with varicocele

ELIGIBILITY:
Inclusion Criteria:

* Infertile men
* Varicocele
* Poor sperm parameters

Exclusion Criteria:

* Men with systemic diseases
* Infertile men due to other causes than varicocele

Ages: 18 Years to 39 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Infertile men with varicocele
Enrollment: 30 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
The Quality of Semen | 6 months
  According to WHO 2010 guidelines regarding semen analysis
  * Sperm concentration (to be more than 15 million sperm per milliliter).
  * Sperm motility (not less than 60% progressive motility).
  * Sperm morphology (not less than 6% normal morphology).

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Benha Faculty of Medecine, Banhā
  - Benha Faculty of Medicine, Banhā

IPD SHARING:
Plan to Share IPD: Undecided